CLINICAL TRIAL: NCT00423657
Title: A Phase 3, Multicenter, Randomized, Double-blind, Comparative Study to Evaluate the Safety and Efficacy of Ceftaroline Versus Vancomycin Plus Aztreonam in Adult Subjects With Complicated Skin and Skin Structure Infection (cSSSI)
Brief Title: Comparative Study of Ceftaroline vs. Vancomycin Plus Aztreonam in Adult Subjects With Complicated Skin Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Senior Vice President, Clinical Development, Cerexa, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P903-07
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Infections
Keywords: Abscess; Antibacterial; Antibiotic; Antimicrobial; Bacterial infection, skin; Ceftaroline; Ceftaroline acetate; Cellulitis; Cephalosporin; Complicated skin and skin structure infection (cSSSI); cSSSI; Intravenous; Methicillin-resistant Staphylococcus Aureus (MRSA); PPI-0903; Prodrug; Skin disease, bacterial; Skin infection; Staphylococcal skin infection; Staphylococcus aureus; Streptococcal skin infection; Surgical site infection; TAK-599
MeSH Terms: conditions — Bacterial Infections; Abscess; Skin Diseases, Bacterial; Cellulitis; Staphylococcal Skin Infections; Staphylococcal Infections; Surgical Wound Infection | interventions — Ceftaroline; Vancomycin; Aztreonam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline fosamil for Injection (Experimental): Ceftaroline fosamil 600 mg administered intravenously over 60 minutes every 12 hours, followed by placebo administered over 60 minutes every 12 hours.
  Interventions: Drug: ceftaroline; Drug: Placebo
- IV Vancomycin plus IV Aztreonam (Active Comparator): Vancomycin 1 g administered over 60 minutes every 12 hours followed by aztreonam 1 g administered over 60 minutes every 12 hours.
  Interventions: Drug: vancomycin plus aztreonam

INTERVENTIONS:
Drug: ceftaroline — 600 mg parenteral infused over 60 minutes, every 12 hours for 5 to 14 days
  Other Names: Experimental
  Arms: Ceftaroline fosamil for Injection
Drug: vancomycin plus aztreonam — vancomycin at 1 g parenteral infused over 60 minutes followed by aztreonam 1 g infused over 60 minutes, every 12 hours, for 5 to 14 days.
  Other Names: Active Comparator
  Arms: IV Vancomycin plus IV Aztreonam
Drug: Placebo — Ceftaroline fosamil 600 mg administered intravenously over 60 minutes every 12 hours, followed by placebo administered over 60 minutes every 12 hours.
  Arms: Ceftaroline fosamil for Injection

SUMMARY:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of complicated skin infections in adults.

DETAILED DESCRIPTION:
Additional purpose of this study is to compare ceftaroline effectivity versus Vancomycin plus Aztreonam in the treatment of complicated skin infections in adults.

ELIGIBILITY:
Inclusion Criteria:

* Skin and skin structure infection (SSSI) that involves deeper soft tissue or requires significant surgical intervention, or cellulitis or abscess on lower extremity which occurs in subjects with diabetes mellitus or well-documented peripheral vascular disease.

Exclusion Criteria:

* Prior treatment of current complicated skin and skin structure infection (cSSSI) with an antimicrobial.
* Failure of vancomycin or aztreonam as therapy for the current cSSSI, or prior isolation of an organism with in vitro resistance to vancomycin or aztreonam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wilcox, MD, Principal Investigator — Old Medical School
Locations (49):
- United States (17):
  - Investigational Site, Buena Park, California
  - Investigational Site, Hawaiian Gardens, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Pasadena, California
  - Investigational Site, San Diego, California
  - Investigational Site, San Jose, California
  - Investigational Site, Atlantis, Florida
  - Investigational Site, Columbus, Georgia
  - Investigational Site, Marietta, Georgia
  - Investigational Site, Springfield, Illinois
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Minneapolis, Minnesota
  - Investigational Site, Butte, Montana
  - Investigational Site, Somers Point, New Jersey
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Tacoma, Washington
  - Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - Investigational Site, Buenos Aires
  - Investigational Site, Córdoba
  - Investigational Site, Santa Fe
- Austria (3):
  - Investigational Site, Braunau am Inn
  - Investigational Site, Graz
  - Investigational Site, Sankt Pölten
- Investigational Site, Sao Paula, Brazil
- Chile (2):
  - Investigational Site, Temuco
  - Investigational Site, Valdivia
- Germany (5):
  - Investigational Site, Cottbus
  - Investigational Site, Dortmund
  - Investigational Site, Homburg/Saar
  - Investigational Site, Mainz
  - Investigational Site, Wiesbaden
- Investigational Site, Riga, Latvia
- Mexico (2):
  - Investigational Site, Guadalajara, Jalisco
  - Investigational Site, Seattle Zapopan, Jalisco
- Poland (7):
  - Investigational Site, Bielsko-Biala
  - Investigational Site, Krakow
  - Investigational Site, Lodz
  - Investigational Site, Lublin
  - Investigational Site, Poznan
  - Investigational Site, Warsaw
  - Investigational Site, Wroclaw
- Russia (3):
  - Investigational Site, Moscow
  - Investigational Site, Moscow Region
  - Investigational Site, Saint Petersburg
- Ukraine (4):
  - Investigational Site, Kharkiv
  - Investigational Site, Kyiv
  - Investigational Site, Lviv
  - Investigational Site, Zaporizhya
- Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Wilcox M, Yan JL, Gonzalez PL, Dryden M, Stone GG, Kantecki M. Impact of Underlying Comorbidities on Outcomes of Patients Treated with Ceftaroline Fosamil for Complicated Skin and Soft Tissue Infections: Pooled Results from Three Phase III Randomized Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):217-230. doi: 10.1007/s40121-021-00557-w. Epub 2021 Nov 6. PMID 34741280
- [Derived] Corey GR, Wilcox MH, Gonzalez J, Jandourek A, Wilson DJ, Friedland HD, Das S, Iaconis J, Dryden M. Ceftaroline fosamil therapy in patients with acute bacterial skin and skin-structure infections with systemic inflammatory signs: A retrospective dose comparison across three pivotal trials. Int J Antimicrob Agents. 2019 Jun;53(6):830-837. doi: 10.1016/j.ijantimicag.2019.01.016. Epub 2019 Feb 1. PMID 30716446
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Corrado ML. Integrated safety summary of CANVAS 1 and 2 trials: Phase III, randomized, double-blind studies evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. J Antimicrob Chemother. 2010 Nov;65 Suppl 4:iv67-iv71. doi: 10.1093/jac/dkq256. PMID 21115456
- [Derived] Wilcox MH, Corey GR, Talbot GH, Thye D, Friedland D, Baculik T; CANVAS 2 investigators. CANVAS 2: the second Phase III, randomized, double-blind study evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. J Antimicrob Chemother. 2010 Nov;65 Suppl 4:iv53-iv65. doi: 10.1093/jac/dkq255. PMID 21115455
- [Derived] Corey GR, Wilcox M, Talbot GH, Friedland HD, Baculik T, Witherell GW, Critchley I, Das AF, Thye D. Integrated analysis of CANVAS 1 and 2: phase 3, multicenter, randomized, double-blind studies to evaluate the safety and efficacy of ceftaroline versus vancomycin plus aztreonam in complicated skin and skin-structure infection. Clin Infect Dis. 2010 Sep 15;51(6):641-50. doi: 10.1086/655827. PMID 20695801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from March 2007 to December 2007
Pre-assignment Details: Patients were screened for up to 24 hours
Groups:
- Ceftaroline for Injection: Ceftaroline fosamil 600 mg administered intravenously over 60 minutes every 12 hours, followed by placebo administered over 60 minutes every 12 hours.
Period: Overall Study
Arm/Group | Ceftaroline for Injection | IV Vancomycin Plus IV Aztreonam
Started | 342 | 338
Completed | 316 | 313
Not Completed | 26 | 25
Not completed — Withdrew consent | 10 | 8
Not completed — Non-compliance | 0 | 1
Not completed — Other | 15 | 16
Not completed — Request of sponsor/investigator | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline for Injection | IV Vancomycin Plus IV Aztreonam | Total
Number analyzed (Participants) | 342 | 338 | 680
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  >18 and < 65 years | 281 | 291 | 572
  >=65 years | 61 | 47 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (16.98) | 47.5 (16.07) | 47.7 (16.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 137 | 255
  Male | 224 | 201 | 425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 59 | 122
  Not Hispanic or Latino | 279 | 279 | 558
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate at Test of Cure (TOC) (MITT Population)
Description: Cure: Total resolution of all signs and symptoms of the baseline infection, or improvement of the infection such that no further antimicrobial therapy was necessary.
  Failure: Requirement of alternative antimicrobial therapy for primary infection of complicated skin and skin structure infection (cSSSI) due to inadequate response, recurrence, new infection at the same site; treatment-limiting adverse event (AE); requirement for surgery due to failure of study drug; diagnosis of osteomyelitis after Study Day 8; or death caused by cSSSI.
  Indeterminate: Inability to determine an outcome
Time Frame: 8-15 days after last dose of study drug administration
Population: MITT (Modified Intent to Treat) - all subjects that received any amount of study drug
Measure: Number; unit: participants
Arm/Group | Ceftaroline for Injection | IV Vancomycin Plus IV Aztreonam
Number analyzed (Participants) | 342 | 338
participants
  Clinical Cure | 291 | 289
  Clinical Failure | 25 | 28
  Indeterminate | 26 | 21
Statistical Analysis 1: Comparison: Ceftaroline for Injection vs IV Vancomycin Plus IV Aztreonam; The primary objective of this study was to determine the noninferiority in clinical cure rate of ceftaroline in comparison with vancomycin plus aztreonam in adult subjects with cSSSI; Test type: Non-Inferiority or Equivalence — A two-sided 95% confidence interval (CI) for the observed difference in the primary outcome measure between ceftaroline and vancomycin plus aztreonam was calculated. Noninferiority was concluded if the lower limit of the 95%CI was higher than -10%; Risk Difference (RD) = -0.4, 95% CI 2-sided [-5.8 to 5.0] — Risk difference corresponds to Ceftaroline clinical cure rate minus Vancomycin plus Aztreonam clinical cure rate. The confidence interval was calculated using the Miettinen and Nurminen method without adjustment

2. Primary Outcome: The Primary Efficacy Outcome Measure Was the Per-subject Clinical Cure Rate at the TOC Visit in the Clinically Evaluable (CE) Populations.
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

3. Secondary Outcome: To Evaluate the Microbiological Success Rate at the TOC Visit
Time Frame: 8-15 days after the last dose of study drug
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate the Clinical Response at the End of Therapy (EOT) Visit
Time Frame: last day of study drug administration
Reporting Status: Not Posted

5. Secondary Outcome: To Evaluate the Clinical and Microbiological Response by Pathogen at the TOC Visit
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

6. Secondary Outcome: To Evaluate Clinical Relapse at the Late Follow Up (LFU) Visit
Time Frame: 21 to 35 days after the last dose of study drug
Reporting Status: Not Posted

7. Secondary Outcome: To Evaluate Microbiological Reinfection or Recurrence at the LFU Visit
Time Frame: 21-35 days after last dose of study drug
Reporting Status: Not Posted

8. Secondary Outcome: To Evaluate Safety
Time Frame: first study drug dose through TOC
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All safety analyses were performed on the Safety Population which consists of all subjects who received any amount of actual study drug.
Arm/Group | Ceftaroline for Injection | IV Vancomycin Plus IV Aztreonam
Serious Adverse Events (participants affected / at risk) | 14/341 | 16/339
Other Adverse Events (participants affected / at risk) | 144/341 | 159/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline for Injection (N=341) | IV Vancomycin Plus IV Aztreonam (N=339)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Central line infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postprocedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline for Injection (N=341) | IV Vancomycin Plus IV Aztreonam (N=339)
Diarrhea (Gastrointestinal disorders) | 22 (22) | 15 (15)
Nausea (Gastrointestinal disorders) | 21 (21) | 19 (19)
Headache (Nervous system disorders) | 18 (18) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (13) | 28 (28)
Insomnia (Psychiatric disorders) | 12 (12) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 10 (10)
Vomiting (Gastrointestinal disorders) | 11 (11) | 9 (9)
Constipation (Gastrointestinal disorders) | 10 (10) | 11 (11)
Hypertension (Vascular disorders) | 8 (8) | 3 (3)
Blood pressure increased (Investigations) | 7 (7) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
Alanine aminotransferase increase (Investigations) | 5 (5) | 7 (7)
Pyrexia (General disorders) | 5 (5) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 8 (8)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No